CLINICAL TRIAL: NCT04774276
Title: Protocol in Reeducation Occupational Therapist in Coronary Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN022021/CHUSTE
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Myocardial Infarction; Coronary Artery Disease
Keywords: occupational therapy; quality of life
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Occupational Therapists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with occupational therapist: Patient with Coronary Artery Disease (CAD) will be included. They will have the cardiac rehabilitation protocol (4 weeks) with occupational therapist as usual practice. The inclusion in this group will be prospective, from January 2021.
  Interventions: Other: cardiac rehabilitation protocol with occupational therapist
- Group without occupational therapist: Patient with Coronary Artery Disease (CAD) will be included. They have done the cardiac rehabilitation protocol (4 weeks) without occupational therapist until december 2020. The inclusion in this group will be retrospective,
  Interventions: Other: cardiac rehabilitation protocol without occupational therapist

INTERVENTIONS:
Other: cardiac rehabilitation protocol without occupational therapist — cardiac rehabilitation protocol without occupational therapist will be performed (usual practice before January 2021).
  Groups: Group without occupational therapist
Other: cardiac rehabilitation protocol with occupational therapist — This intervention (occupational therapist) have been added since 2021 for all patients who need a cardiac rehabilitation protocol.
  Occupational therapy is scheduled with sessions 3 times a week for 1 month.
  Groups: Group with occupational therapist

SUMMARY:
The quality of life, linked to physical, social and mental performance in people with coronary heart disease represents the primary goals in terms of rehabilitation. This is often developed to meet the expected performance standard in order to give the person effective autonomy. However, is the occupational balance always evaluated? and this management adapted? Does occupational therapist, expert in autonomy and independence in multiple illnesses and disabilities, has a major role to play in cardiac rehabilitation? This area of expertise and the application of occupational therapy to coronary patients seems appropriate, if not necessary. However, there are few scientific studies on the need to include occupational therapy within cardiac rehabilitation protocols.

DETAILED DESCRIPTION:
The occupational therapy goals are in line with the theoretical objectives of coronary rehabilitation. At present, there is a lack of data on the benefits of coronary occupational therapy rehabilitation.

Goals : Evaluation of the quality of life of coronary heart patients who have benefited from cardiac rehabilitation optimized by secondary occupational therapy sessions:

Evaluation of aerobic and anaerobic performance of coronary heart patients who have benefited from cardiac rehabilitation optimized by occupational therapy sessions.

Evaluation of aerobic and anaerobic performance of coronary heart patients who have benefited from cardiac rehabilitation optimized by occupational therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Included in the cardiac rehabilitation protocol in Saint Etienne university hospital

Exclusion Criteria:

* Patients who not perform all sessions of the cardiac rehabilitation protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease (CAD) needed a cardiac rehabilitation protocol
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Short Form (SF-36) questionnaire score | week 5
  The SF-36 is a self-questionnaire to assess the quality of life and contains 36 items with minimum score 0 (bad quality life) and maximum score at 100 (good quality life).
  Done one week after the end of cardiac rehabilitation protocol

SECONDARY OUTCOMES:
Strength of biceps muscle (Kg) | week 5
  Measured by handgrip
  Done one week after the end of cardiac rehabilitation protocol

OTHER OUTCOMES:
6 minutes walk test (TM6) | week 5
  Measured by the distance in metres at the walking time of 6 minutes.
  Done one week after the end of cardiac rehabilitation protocol

CONTACTS AND LOCATIONS:
Overall Officials: DAVID HUPIN, MD, Principal Investigator — CHU ST ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No